CLINICAL TRIAL: NCT06200077
Title: Clinical Outcomes of Different Staged Ridge-Splitting Techniques Using Piezo-Electric Surgery in Atrophic Posterior Mandible
Brief Title: Patient Outcomes of Staged Ridge-splitting Using Piezo-electric Surgery in Atrophic Posterior Mandible
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A01051021
Record Dates: First submitted 2023-12-28; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2021-11

CONDITIONS: Alveolar Ridge Augmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Ridge-Splitting Group (Sham Comparator): Six dental implant sites were prepared in three patients initially through ridge splitting technique associated with bone grafting followed by implants insertion after 4 months later.
  Interventions: Procedure: Modified Ridge-Splitting
- Modified 3-Staged Ridge-Splitting Group (Active Comparator): Six dental implant sites were prepared in four patients through mucogingival and bony incision initially then after 3-4 weeks ridge splitting with bone grafting were done, followed by implants insertion after 4 months later.
  Interventions: Procedure: Modified Ridge-Splitting
- Modified 2-Staged Ridge-Splitting Group (Experimental): Six dental implant sites were prepared in three patients initially through mucogingival, and bony incision followed by ridge splitting technique, bone grafting and implants insertion at the same time after 4 weeks from the bony incision.
  Interventions: Procedure: Modified Ridge-Splitting

INTERVENTIONS:
Procedure: Modified Ridge-Splitting — Unlike the conventional ridge-splitting where bone grafting is done in the same visit after ridge splitting, modified ridge splitting involves splitting the ridge only at the first visit, then bone grafting is done either alone afterwards in the second visit (Modified 3-Staged Ridge-Splitting Group) and dental implants will be placed in the third visit, or, as in the Modified 2-Staged Ridge-Splitting Group, bone grafting and dental implants placement will be done in the second visit.

SUMMARY:
This study aims to evaluate the clinical and radiographic outcomes of different staged ridge-splitting techniques for management of severely resorbed lower jaws in the posterior region. The study is designed as a clinical trial, so that three different interventions would be compared for a conclusion highlighting the relative best of them.

DETAILED DESCRIPTION:
In the context of the care of severely resorbed lower jaws in the posterior region, the purpose of this study is to evaluate the clinical and radiographic outcomes of several stepwise ridge-splitting procedures. The study is supposed to be a clinical trial, with the purpose of comparing three distinct therapies in order to get a result that highlights which of them is the most effective in comparison to the others.

ELIGIBILITY:
Inclusion Criteria:

* Patients were free from any relevant systemic diseases according to American society of Anesthesiologists classifications.
* Patients of single or multiple missing teeth in the posterior mandible.
* A ridge width of minimum 4mm and a 10 mm ridge height with 2mm minimum above Inferior Alveolar Nerve (IAN) were present in CBCT images.
* Absence of buccal concavities at the planned implant site.

Exclusion Criteria:

* History of any systemic diseases or medication that alters bone metabolism.
* Poor oral hygiene.
* Heavy smoker (more than 20 cigarettes/day) or alcoholic patients.
* Chemotherapy or radiation therapy to the head and neck region in the last 12 months prior to the proposed implant therapy.
* Patients currently on or with a history of bisphosphonate therapy.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Alveolar ridge width | immediately after implant placement, immediately after implant loading and six months after implant loading
  Radiographically via Cone-beam Computed Tomography (CBCT), the width of the alveolar bone was measured horizontally from the buccal to lingual cortex below the crest of the alveolar bone from 3 levels at 1 mm, 3 mm and 6 mm on three cross-sections by the CBCT software (OnDemand, Cybermed Inc, Korea).

SECONDARY OUTCOMES:
Implant stability | immediately after implant placement, immediately after implant loading and six months after implant loading
  Smartpeg was installed in the dental implant fixture. From both buccal and lingual directions, an analyzer probe was located closer to the Smartpeg, and the implant stability quotient (ISQ) values were obtained from the Osstell Monitor

CONTACTS AND LOCATIONS:
Overall Officials: Mena Tamer, MSc, Principal Investigator — Faculty of Dentistry, Mansoura University
Locations (1):
- Faculty of Dentistry, Mansoura University, Al Mansurah, Dakahlyia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hu GH, Froum SJ, Alodadi A, Nose F, Yu YP, Suzuki T, Cho SC. A Three-Stage Split-Crest Technique: Case Series of Horizontal Ridge Augmentation in the Atrophic Posterior Mandible. Int J Periodontics Restorative Dent. 2018 July/August;38(4):565-573. doi: 10.11607/prd.2907. Epub 2018 Mar 13. PMID 29534117